CLINICAL TRIAL: NCT03758183
Title: Cost Effectiveness of Two-stage Algorithm (Prolotherapy Injections Prior to Total Knee Arthroplasty) in the Management of Advanced Stage Knee Osteoarthritis
Brief Title: Cost Effectiveness of Prolotherapy Injections Prior to Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Tokat State Hospital (Other Government)
Responsible Party: Principal Investigator, Serkan Akpancar, Dr, Tokat State Hospital
Other Study IDs: TokatSH
Record Dates: First submitted 2018-11-08; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty; Prolotherapy; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Injections; Prolotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- two-stage algorithm: Prolotherapy injections (PrT) combined with rehabilitation protocol (RP) prior to total knee arthroplasty (TKA)
  Interventions: Procedure: total knee arthroplasty
- one-stage algorithm: total knee arthroplasty (TKA)
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty
  Other Names: injection; prolotherapy

SUMMARY:
This study compared the cost effectiveness of two-stage algorithm (prolotherapy injections (PrT) combined with rehabilitation protocol (RP) prior to total knee arthroplasty (TKA)) and one-stage algorithm (TKA) in the management of advanced stage knee osteoarthritis.

DETAILED DESCRIPTION:
The aim of the present study was to compare the cost effectiveness of two-stage algorithm (prolotherapy injections (PrT) combined with rehabilitation protocol (RP) prior to total knee arthroplasty (TKA)) and one-stage algorithm (TKA) in the management of advanced stage knee osteoarthritis.

A total of 197 patients who had chronic knee osteoarthritis were included in the present study. The patients were divided into two groups as two-stage algorithm (PrT combined with RP prior to TKA), (Group A, n=98) and one-stage (TKA),(Group B, n=99). Clinical effectiveness was evaluated via Visual Analog Scale (VAS), The Western Ontario and McMaster Universities Arthritis Index (WOMAC) at baseline and 3-, 6-, 12-, and 18-month follow-ups. Utility scores of the groups were obtained by extracting and converting WOMAC scores to health utilities index mark 3 scores. Cost-utility per quality-adjusted life years (QALY) and Incremental cost-effectiveness ratios (ICERs) of each group were calculated.

ELIGIBILITY:
Inclusion Criteria:

* III and IV levels of knee osteoarthritis according to Kellgren-Lawrence
* Had at least six months of symptoms resistant to at least three months of conservative methods (lifestyle modification, weight reduction, regular exercise, physiotherapy, non-steroidal anti-inflammatory drugs, intraarticular injection methods) -

Exclusion Criteria:

* With rheumatic diseases, immune diseases or other systemic inflammatory diseases
* With active infection, osteomyelitis or history of chronic infection around knee joint
* Had undergone previous operation on knee
* Had bleeding tendency (hereditary or acquired)
* Pregnant patients

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age of the patients varied between 50 and 90
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 18 months
  Self reported pain intensity. Each item is scored 0-10 (0=no pain; 10= pain as bad as can be), yielding a total between 0 and 10.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 18 months
  Self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. Each item is scored 0-96 (0=minimum; 96= as bad as can be), yielding a total between 0 and 96.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Akpancar, Dr, Study Director — Tokat State Hospital
Locations (1):
- Serkan Akpancar, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All primary and secondary data will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available with in 3 months of the study completed
Access Criteria: Data will be reviewed by external independent review panel. Requesters will be required to sign a data access agreement.